CLINICAL TRIAL: NCT00673894
Title: Study of the Effects of Glutamine on Glycemia, Glucagon-like Peptide-1 (GLP-1) and Insulin Secretion in Man
Brief Title: Effects of Glutamine on GLP-1 and Insulin Secretion in Man
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Dr Jerry Greenfield, Prof, Garvan Institute of Medical Research
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H07/059
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glutamine+Sitagliptin (Experimental): Glutamine 30 g/d (15 g with breakfast and dinner) + Sitagliptin
  Interventions: Drug: Sitagliptin
- Glutamine+Placebo (Placebo Comparator): Glutamine 30 g/d (15 g with breakfast and dinner) + placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Glutamine 30g +sitagliptin 100mg
  Other Names: Januvia
  Arms: Glutamine+Sitagliptin
Drug: Placebo — Glutamine 30g +placebo (matching sitagliptin 100 mg)
  Arms: Glutamine+Placebo

SUMMARY:
This study investigated the effect of glutamine, an amino acid, glycemia, glucagon-like peptide-1 (GLP-1) and insulin in participants with type 2 diabetes.

DETAILED DESCRIPTION:
In this study, we investigated the effect of glutamine, an amino acid, on glycemia and on GLP-1 and insulin in participants with type 2 diabetes. Preliminary data published by our group suggests that glutamine is a strong determinant of GLP-1 secretion in vitro. We tested the hypothesis that glutamine lowers postprandial blood glucose and investigated whether the dipeptidyl peptidase-4 (DPP-4) inhibitor sitagliptin modifies this effect.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, on metformin or diet alone (not sulphonylureas or insulin)

Exclusion Criteria:

* Malabsorption, renal or liver disease, treatment with steroids

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry R Greenfield, MD, PhD, Principal Investigator — Garvan Institute of Medical Research
Locations (1):
- Clinical Research Facility, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Samocha-Bonet D, Wong O, Synnott EL, Piyaratna N, Douglas A, Gribble FM, Holst JJ, Chisholm DJ, Greenfield JR. Glutamine reduces postprandial glycemia and augments the glucagon-like peptide-1 response in type 2 diabetes patients. J Nutr. 2011 Jul;141(7):1233-8. doi: 10.3945/jn.111.139824. Epub 2011 May 18. PMID 21593352
- [Result] Samocha-Bonet D, Chisholm DJ, Holst JJ, Greenfield JR. L-glutamine and whole protein restore first-phase insulin response and increase glucagon-like peptide-1 in type 2 diabetes patients. Nutrients. 2015 Mar 24;7(4):2101-8. doi: 10.3390/nu7042101. PMID 25811109
- [Result] Samocha-Bonet D, Chisholm DJ, Gribble FM, Coster AC, Carpenter KH, Jones GR, Holst JJ, Greenfield JR. Glycemic effects and safety of L-Glutamine supplementation with or without sitagliptin in type 2 diabetes patients-a randomized study. PLoS One. 2014 Nov 20;9(11):e113366. doi: 10.1371/journal.pone.0113366. eCollection 2014. PMID 25412338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 of 22 participants were randomized. Of those not randomized, 7 did not meet the inclusion criteria
Groups:
- Sitagliptin, Then Placebo: Participants first received Glutamine 30 g/d + Sitagliptin (100 mg/d) for 4 weeks. After a washout period of 4-6 weeks, they then received Glutamine 30 g/d + Placebo (matching Sitagliptin 100 mg) for 4 weeks
- Placebo, Then Sitagliptin: Participants first received Glutamine 30 g/d + Placebo (matching Sitagliptin 100 mg) for 4 weeks. After a washout period of 4-6 weeks, they then received Glutamine 30 g/d + Sitagliptin (100 mg/d) for 4 weeks
Period: First Intervention 4 Weeks
Arm/Group | Sitagliptin, Then Placebo | Placebo, Then Sitagliptin
Started (First Intervention Duration 4 weeks) | 8 | 7
Completed | 6 | 7
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout 4-6 Weeks
Arm/Group | Sitagliptin, Then Placebo | Placebo, Then Sitagliptin
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Second Intervention 4 Weeks
Arm/Group | Sitagliptin, Then Placebo | Placebo, Then Sitagliptin
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized to receive either sitagliptin 100 mg tablet or placebo tablet (matching sitagliptin 100 mg)
Groups:
- First Received Sitagliptin, Then Placebo: Participants first received Glutamine 30 g/d + Sitagliptin (100 mg/d) for 4 weeks. After a washout period of 4-6 weeks, they then received Glutamine 30 g/d + Placebo (matching Sitagliptin 100 mg) for 4 weeks
- First Received Placebo, Then Sitagliptin: Participants first received Glutamine 30 g/d + Placebo (matching Sitagliptin 100 mg/d) for 4 weeks. After a washout period of 4-6 weeks, they then received Glutamine 30 g/d +Sitagliptin (100 mg) for 4 weeks
- Total: Total of all reporting groups
Arm/Group | First Received Sitagliptin, Then Placebo | First Received Placebo, Then Sitagliptin | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 individuals withdrew from the study
  Participants
    number analyzed (Participants) | 6 | 7 | 13
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 6
    >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 individuals withdrew
  years
    number analyzed (Participants) | 6 | 7 | 13
    (all) | 64 (8) | 65 (5) | 65 (6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 individuals withdrew from the study
  Participants
    number analyzed (Participants) | 6 | 7 | 13
    Female | 2 | 2 | 4
    Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants] — Population: 2 participants withdrew
  participants
    Australia: number analyzed (Participants) | 6 | 7 | 13
    Australia | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glucose Area Under the Curve (AUC)
Description: The area under the curve (AUC) of the postprandial glucose following a meal challenge
Time Frame: 0 to 180 minutes
Population: The primary aim of this randomized crossover study was to determine the glycemic effect of 4 weeks of glutamine (15 bd) supplementation with sitagliptin (100 mg/d) or placebo in type 2 diabetes patients treated with metformin.
Measure: Mean (Standard Deviation); unit: mmol/L*t
Groups:
- Glutamine+Placebo: Glutamine 30 g/d (15 g with breakfast and dinner) + placebo
  Placebo: Glutamine 30g +placebo
Arm/Group | Glutamine+Sitagliptin | Glutamine+Placebo
Number analyzed (Participants) | 13 | 13
mmol/L*t | 1341 (180) | 1463 (179)

2. Secondary Outcome: Fructosamine
Description: The blood concentration of the glycemic control marker fructosamine
Time Frame: 4 weeks
Population: The secondary aim of this randomized crossover study was to determine the glycemic effect of 4 weeks of glutamine (15 bd) supplementation with sitagliptin (100 mg/d) or placebo in type 2 diabetes patients treated with metformin.
Measure: Mean (Standard Deviation); unit: micro mol per litre
Arm/Group | Glutamine+Sitagliptin | Glutamine+Placebo
Number analyzed (Participants) | 13 | 13
micro mol per litre | 244 (41) | 240 (30)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 4 weeks treatment with the first arm and then during the 4 weeks of treatment with the second arm. Total of 8 weeks.
Description: Adverse events were collected during physical visits to the Clinical Research Facility at the Garvan Institute of Medical Research. Participants were interviewed by the Study Nurse and asked to report any event or symptom they experienced during each of the 4 weeks treatments.
Groups:
- Sitagliptin: Glutamine 30 g/d (15 g with breakfast and dinner) + Sitagliptin
- Placebo: Glutamine 30 g/d (15 g with breakfast and dinner) + Placebo
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes